CLINICAL TRIAL: NCT01566578
Title: A Physiological Study on Downregulation of EGF-receptors in the Skin by Topical Exposition With EGF
Acronym: EGFR
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ennar Pharmaceuticals AF (Industry)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EGFR-Study
Record Dates: First submitted 2012-03-21; First posted 2012-03-29 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-08

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EGF Cream (Experimental)
  Interventions: Drug: Human recombinant epidermal growth factor
- Placebo cream (Placebo Comparator)
  Interventions: Other: Placebo cream

INTERVENTIONS:
Drug: Human recombinant epidermal growth factor — topical
  Arms: EGF Cream
Other: Placebo cream — Dermal cream without EGF
  Arms: Placebo cream

SUMMARY:
Investigation of EGF-Receptor Downregulation by topical EGF (dermal cream) exposition.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Mild to moderate psoriasis (all types) with active plaques on both body sides accessible for biopsy and self product application
* EGFR immunohistochemistry score > 5
* Male
* Age 18-60 years

Exclusion Criteria:

* Systemic psoriasis treatment 3 months prior and during the study
* Local psoriasis treatment on the investigational sites in the last 30 days or during the study
* Known hypersensitivity or allergy to the EGF containing product (Newskin) and/or to Vaseline/10% salicylic acid and/or to local anaesthetics of the amid type
* Known or suspected non-compliance to study protocol Coagulopathy or treatment with anticoagulants
* History of malignant disease Other clinically relevant concomitant disease state Participation in another investigational drug study in the last 30 days

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in EGFR density in epidermis of psoriasis lesion | Day 66
  Punch biopsies of the treated psoriasis lesion will be performed before study treatment start (day 7) and at the end of the treatment, which is on day 66.
  EGFR immunohistochemistry will be performed with a murine antibody directed against the extracellular domain of human EGFR. A pathologist blinded to the patient's characteristics and treatment modalities assesses the immunohistochemistry staining in three epidermal layers. A score ranging form 0 (no staining) to 3 (intense staining) is applied, resulting in a total score ranging form 0 (3x0) to 9 (3x3).

SECONDARY OUTCOMES:
Change to baseline in target lesion severity score (PASI) | Day 80
  A blinded dermatologist assesses the treated psoriasis plaque clinically using the lesion assessment part of the PASI score, assessing 3 qualities (thicknes, redness and scaling) of the lesion. Score ranges from 0 (absent) to 4 (very severe), resulting in a total score of 0 to 12 (3 x 4)
Change to baseline in histological feature: thickness of the epidermis | Day 66
  Punch biopsies of the treated psoriasis lesion will be performed before study treatment start (day 7) and at the end of the treatment on day 66.
  A pathologist blinded to the patient's characteristics and treatment modalities assesses the following histological features: thicknes of the epidermis, acanthosis and epidermal/dermal lymphocytic infiltrates. Each characteristic is scored as follows: 0 = normal, + = mild, and ++ = marked.
Number of participants with adverse events | Day 80
  At every visit the patients are asked about the occurence of adverse events. The last visit is on day 80. All adverse events will be recorded in the crf.
Change to baseline in the histological feature: acanthosis | Day 66
  Punch biopsies of the treated psoriasis lesion will be performed before study treatment start (day 7) and at the end of the treatment on day 66.
  A pathologist blinded to the patient's characteristics and treatment modalities assesses the following histological features: thicknes of the epidermis, acanthosis and epidermal/dermal lymphocytic infiltrates. Each characteristic is scored as follows: 0 = normal, + = mild, and ++ = marked.
Change to baseline in histological feature: epidermal/dermal lymphocytic infiltrates | Day 66
  Punch biopsies of the treated psoriasis lesion will be performed before study treatment start (day 7) and at the end of the treatment on day 66.
  A pathologist blinded to the patient's characteristics and treatment modalities assesses the following histological features: thicknes of the epidermis, acanthosis and epidermal/dermal lymphocytic infiltrates. Each characteristic is scored as follows: 0 = normal, + = mild, and ++ = marked.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kündig, MD, Principal Investigator — University Hospital Zurich, Dermatology Clinic
Locations (1):
- University Hospital Zurich, Dermatology Clinic, Zurich, Canton of Zurich, Switzerland